CLINICAL TRIAL: NCT03698591
Title: Testing a Neurocognitive Model of Distancing Using Transcranial Magnetic Stimulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00100171
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Emotion Regulation; Real Versus Sham Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the lead experimenter nor the subject will know which arm they will complete first. The secondary experimenter will use a randomized counter-balanced log to determine the order of sequences will take place. The secondary experimenter will set up the device while the lead experimenter is out of the room to preserve blindness to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial magnetic stimulation (TMS), then Sham TMS. (Experimental): Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task. Thirty minutes after stimulation, experimenters will employ a sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.
  Interventions: Device: Transcranial magnetic stimulation task
- Sham TMS, then Transcranial magnetic stimulation (TMS) (Sham Comparator): Experimenters will employ a sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject. Experimenters have defined the target coordinates for the stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task. Thirty minutes post sham stimulation, experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates.
  Interventions: Device: Sham transcranial magnetic stimulation task

INTERVENTIONS:
Device: Transcranial magnetic stimulation task — Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task.
  Other Names: TMS
  Arms: Transcranial magnetic stimulation (TMS), then Sham TMS.
Device: Sham transcranial magnetic stimulation task — A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.
  Other Names: Sham TMS
  Arms: Sham TMS, then Transcranial magnetic stimulation (TMS)

SUMMARY:
Distancing oneself from a current distressing situation is a mental skill that can help people to manage their emotions. However, little is known about how distancing works in the brain. Recently developed tools in neuroscience that can modify brain activity might be able to make distancing more or less effective. In doing so, the results could lead to a better understanding of the cognitive processes and neural circuits that support distancing as a form of emotion regulation. If successful, this research may lead to the development of new treatments to help those who suffer from stress-related disorders, such as anxiety and depression.

DETAILED DESCRIPTION:
Distancing is an emotion regulation skill that relies in part on self-projection, or the ability to shift perspective from the here and now to a simulated time, place, or person. Based on prior review and meta-analysis of the distancing literature, a new model has been developed of the neurocognitive processes that support distancing. The proposed experiment will test the model causally through a neural intervention that should impair or enhance the ability of healthy adults to successfully apply distancing to down-regulate negative affect. In the model, it is hypothesized that the temporoparietal junction (TPJ) was a key region mediating the self-projection aspect of distancing. Leveraging recent functional magnetic resonance imaging (fMRI) work, the experiment will functionally modulate this region through inhibitory transcranial magnetic stimulation (TMS) to test its causal role in distancing. Importantly, the proposed work shifts emphasis from traditional models of emotion regulation, which implicate frontal executive control mechanisms, to new cognitive processes and brain targets that can ultimately lead to novel approaches to treat affective disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-39 years inclusive
* Willing to provide informed consent
* English speaking
* Signed HIPAA authorization

Exclusion Criteria:

* Current or recent (within the past 6 months) substance abuse or dependence, excluding nicotine and caffeine (assessed via urine test).
* Current serious medical illness (assessed via self report).
* History of seizure except those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain surgery, head injury, cranial metal implants, known structural brain lesion, devices that may be affected by TMS or MRI (pacemaker, medication pump, cochlear implant, implanted brain stimulator) [assessed via TMS Adult Safety Screening form].
* Subjects are unable or unwilling to give informed consent.
* Diagnosed any Axis I Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) disorder (assessed via self report).
* Subjects with a clinically defined neurological disorder (assessed via self report) including, but not limited to:

  1. Any condition likely to be associated with increased intracranial pressure
  2. Space occupying brain lesion.
  3. History of stroke.
  4. Transient ischemic attack within two years.
  5. Cerebral aneurysm.
  6. Dementia.
  7. Parkinson's disease.
  8. Huntington's disease.
  9. Multiple sclerosis.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold (assess via self report).
* Subjects not willing to tolerate the confinement associated with being in the MRI scanner.
* Women who are pregnant or breast-feeding (assessed via urine test).
* Blindness.
* Inability to read or understand English.
* Intracranial implants, such as:

  1. Cochlear implants;
  2. Aneurysms clips;
  3. Shunts;
  4. Stimulators;
  5. Electrodes;
  6. Cardiac pacemakers;
  7. Vagus Nerve stimulation devices.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S LaBar, PhD, Principal Investigator — Duke University Faculty
Locations (1):
- LaBar Lab, Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data relating to the primary and secondary outcomes will be uploaded upon completion of the study.

REFERENCES:
- [Background] Dorfel D, Lamke JP, Hummel F, Wagner U, Erk S, Walter H. Common and differential neural networks of emotion regulation by Detachment, Reinterpretation, Distraction, and Expressive Suppression: a comparative fMRI investigation. Neuroimage. 2014 Nov 1;101:298-309. doi: 10.1016/j.neuroimage.2014.06.051. Epub 2014 Jun 30. PMID 24993897
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Madore KP, Thakral PP, Beaty RE, Addis DR, Schacter DL. Neural Mechanisms of Episodic Retrieval Support Divergent Creative Thinking. Cereb Cortex. 2019 Jan 1;29(1):150-166. doi: 10.1093/cercor/bhx312. PMID 29161358
- [Background] McRae K, Hughes B, Chopra S, Gabrieli JD, Gross JJ, Ochsner KN. The neural bases of distraction and reappraisal. J Cogn Neurosci. 2010 Feb;22(2):248-62. doi: 10.1162/jocn.2009.21243. PMID 19400679
- [Background] Winecoff A, Labar KS, Madden DJ, Cabeza R, Huettel SA. Cognitive and neural contributors to emotion regulation in aging. Soc Cogn Affect Neurosci. 2011 Apr;6(2):165-76. doi: 10.1093/scan/nsq030. Epub 2010 Apr 12. PMID 20385663
- [Derived] Powers JP, Davis SW, Neacsiu AD, Beynel L, Appelbaum LG, LaBar KS. Examining the Role of Lateral Parietal Cortex in Emotional Distancing Using TMS. Cogn Affect Behav Neurosci. 2020 Oct;20(5):1090-1102. doi: 10.3758/s13415-020-00821-5. PMID 32839957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11/1/18 until 5/17/19. Subjects were recruited and screened from the Duke University Brain Imaging Analysis Center (BIAC) research participant pool as well as from e-flyers on Duke University's electronic community bulletin board (DukeList).
Groups:
- Transcranial Magnetic Stimulation (TMS), Then Sham TMS: Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task. Thirty minutes post stimulation, experimenters will employ a sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.
- Sham TMS, Then Transcranial Magnetic Stimulation (TMS): Sham transcranial magnetic stimulation task: A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject. Thirty minutes post sham stimulation, experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation (TMS), Then Sham TMS | Sham TMS, Then Transcranial Magnetic Stimulation (TMS)
Started | 20 | 20
Completed | 15 | 15
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Failed drug screen | 1 | 1
Not completed — Failed health screen | 0 | 1
Not completed — Ineligible for financial compensation | 1 | 0
Not completed — Equipment Error | 1 | 0
Not completed — Could not establish TMS dosage | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who completed the study protocol.
Groups:
- Transcranial Magnetic Stimulation (TMS), Then Sham TMS: Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task. Thirty minutes post stimulation, experimenters will employ a A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.
- Sham TMS, Then Transcranial Magnetic Stimulation: A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task. Thirty minutes post stimulation, experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates.
- Total: Total of all reporting groups
Arm/Group | Transcranial Magnetic Stimulation (TMS), Then Sham TMS | Sham TMS, Then Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 3 | 7 | 10
  Unknown/unlisted | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Valence (Distancing) From Baseline to 30 Minutes Post Stimulation.
Description: Valence is how positive or negative a subject feels. Subjects will be asked to rate how they feel on a 7 point Likert scale ranging from 1 (very negative) to 7 (very positive) after using an emotion regulation technique (distancing) when shown graphic stimuli.
Time Frame: baseline, 30 minutes post stimulation
Population: All subjects who completed the study protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Transcranial Magnetic Stimulation (TMS): Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task.
  Transcranial magnetic stimulation task: Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task.
- Sham TMS: A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.
  Sham transcranial magnetic stimulation task: A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham TMS
Number analyzed (Participants) | 30 | 30
score on a scale | .662 (.565) | .668 (.561)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; The null hypothesis was that distancing performance would not differ by arm of the study. Within-subjects factors included task condition (distancing vs. distraction) and study arm. Study arm order was used as a between-subjects factor; Test type: Other; p = .019, ANOVA — P-value corresponds to 3 way interaction. A priori significance threshold of p < .05; F-statistic = 6.155
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; This analysis evaluated the two-way interaction of task condition and study period. The null hypothesis was that distancing performance would not differ by study period. Within-subjects factors included task condition and study period; Test type: Other; p = .021, ANOVA — P-value corresponds to two-way interaction. A priori significance threshold of p < .05; F-statistic = 5.911
Statistical Analysis 3: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; A dependent-samples t-test was used to compare distancing performance between study periods 1 and 2. The null hypothesis was that distancing performance would not differ by study period; Test type: Other; p = .108, t-test, 2 sided — A priori significance threshold of p < .05; t-statistic = -1.656
Statistical Analysis 4: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; For this analysis, study arm and task condition were used as within-subjects factors, study arm order was used as a between-subjects factor, and TMS stimulator intensity and brain-target-to-scalp distance were used as covariates; Test type: Other; p = .948, ANOVA — A priori threshold of p < .05. This value reflects the test of the main effect of study arm; F-statistic = .004

2. Secondary Outcome: Change in Self-reported Effort (Distancing) From Baseline to 30 Minutes Post Stimulation.
Description: Effort is how difficult it was for a subject to use a specific emotion regulation technique. Subjects will be asked to rate how much effort they felt they used on a 7 point Likert scale ranging from 1 (very little effort) to 7 (very high effort) after using an emotion regulation technique (distancing) when shown graphic stimuli.
Time Frame: baseline, 30 minutes post stimulation
Population: All subjects who completed the study protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham TMS
Number analyzed (Participants) | 30 | 30
score on a scale | 3.610 (.841) | 3.546 (.959)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; The null hypothesis was that distancing self-reported effort would not differ by arm of the study. Within-subjects factors included task condition (distancing vs. distraction) and study arm. Study arm order was used as a between-subjects factor; Test type: Other; p = .862, ANOVA — P-value corresponds to the two way interaction of task condition and study arm . A priori significance threshold of p < .05; F-statistic = .031
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; A follow-up ANOVA was run with within-subjects factors of task condition and study period; Test type: Other; p = .054, ANOVA — P-value corresponds to the main effect of study period. A priori threshold of p < .05; F-statistic = 4.040
Statistical Analysis 3: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; A follow-up dependent-samples t-test was run to test a potential effect of study period on distancing effort; Test type: Other; p = .012, t-test, 2 sided — A priori significance threshold of p < .05; t-statistic = 2.694
Statistical Analysis 4: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; Post-hoc analyses were used to explore treatment effects using covariates related to the treatment parameters. For this analysis, study arm and task condition were used as within-subjects factors, study arm order was used as a between-subjects factor, and TMS stimulator intensity and brain-target-to-scalp distance were used as covariates; Test type: Other; p = .085, ANOVA — A priori threshold of p < .05. This value reflects the test of the main effect of study arm; F-statistic = 3.196
Statistical Analysis 5: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; This analysis examined the effect of study arm specifically on distancing effort. The within-subjects factor was study arm, between-subjects factor was study arm order, and TMS stimulator intensity and brain-target-to-scalp distance were used as covariates; Test type: Other; p = .013, ANOVA — A priori threshold of p < .05. This value reflects the test of the main effect of study arm; F-statistic = 7.162

3. Other Pre Specified Outcome: Change in Self-reported Valence (Distraction) From Baseline to 30 Minutes Post Stimulation.
Description: Valence is how positive or negative a subject feels. Subjects will be asked to rate how they feel on a 7 point Likert scale ranging from 1 (very negative) to 7 (very positive) after using an emotion regulation technique (distraction) when shown graphic stimuli.
Time Frame: baseline, 30 minutes post stimulation
Population: All subjects who completed the study protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham TMS
Number analyzed (Participants) | 30 | 30
score on a scale | .617 (.608) | .710 (.661)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; The null hypothesis was that distraction performance would not differ by arm of the study. Within-subjects factors included task condition (distancing vs. distraction) and study arm. Study arm order was used as a between-subjects factor; Test type: Other; p = .019, ANOVA — P-value corresponds to 3 way interaction. A priori significance threshold of p < .05; F-statistic = 6.155
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; This analysis evaluated the two-way interaction of task condition and study period. The null hypothesis was that distraction performance would not differ by study period. Within-subjects factors included task condition and study period; Test type: Other; p = .021, ANOVA — P-value corresponds to two-way interaction. A priori significance threshold of p < .05; F-statistic = 5.911
Statistical Analysis 3: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; A dependent-samples t-test was used to compare distraction performance between study periods 1 and 2. The null hypothesis was that distraction performance would not differ by study period; Test type: Other; p = .210, t-test, 2 sided — A priori significance threshold of p < .05; t-statistic = 1.282
Statistical Analysis 4: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = .948, ANOVA — A priori threshold of p < .05. This value reflects the test of the main effect of study arm; F-statistic = .004

4. Other Pre Specified Outcome: Change in Self-reported Effort (Distraction) From Baseline to 30 Minutes Post Stimulation.
Description: Effort is how difficult is was for a subject to use a specific emotion regulation technique. Subjects will be asked to rate how much effort they felt they used on a 7 point Likert scale ranging from 1 (very little effort) to 7 (very high effort) after using an emotion regulation technique (distraction) when shown graphic stimuli.
Time Frame: baseline, 30 minutes post stimulation
Population: All subjects who completed the study protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham TMS
Number analyzed (Participants) | 30 | 30
score on a scale | 3.620 (1.083) | 3.590 (1.146)
Statistical Analysis 1: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; The null hypothesis was that distraction self-reported effort would not differ by arm of the study. Within-subjects factors included task condition (distancing vs. distraction) and study arm. Study arm order was used as a between-subjects factor; Test type: Other; p = .862, ANOVA — [p-value comment as in outcome 2, analysis 1]; F-statistic = .031
Statistical Analysis 2: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; A follow-up ANOVA was run with within-subjects factors of task condition and study period; Test type: Other; p = .054, ANOVA — P-value corresponds to the main effect of study period. A priori threshold of p < .05; F-statistic = 4.040
Statistical Analysis 3: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; A follow-up dependent-samples t-test was run to test the effect of study period on distraction effort; Test type: Other; p = .415, t-test, 2 sided — A priori significance threshold of p < .05; t-statistic = .828
Statistical Analysis 4: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; [analysis description as in outcome 2, analysis 4]; Test type: Other; p = .085, ANOVA — A priori threshold of p < .05. This value reflects the test of the main effect of study arm; F-statistic = 3.196
Statistical Analysis 5: Comparison: Transcranial Magnetic Stimulation (TMS) vs Sham TMS; This analysis examined the effect of study arm specifically on distraction performance. The within-subjects factor was study arm, between-subjects factor was study arm order, and TMS stimulator intensity and brain-target-to-scalp distance were used as covariates; Test type: Other; p = .535, ANOVA — A priori threshold of p < .05. This value reflects the test of the main effect of study arm; F-statistic = .396

ADVERSE EVENTS:
Time Frame: 30 minutes
Groups:
- Transcranial Magnetic Stimulation (TMS): Experimenters will employ a continuous theta-burst stimulation (cTBS) sequence using a figure-8 coil positioned tangentially to the scalp over the target coordinates. Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task.
- Sham TMS: A sham version of the TMS intervention where subjects will receive a small electrical stimulation on the scalp via two small electrodes in conjunction with a TMS coil activation. The TMS coil will be reoriented to stimulate into the air away from the scalp, simulating traditional TMS, without inducing any current to the subject.Experimenters have defined the target coordinates for stimulation (Montreal Neuroscience Institute coordinates -53, -53, 23) based on peak objective distancing activation in the left temporal parietal junction (TPJ) in previous fMRI studies using the same task.
Arm/Group | Transcranial Magnetic Stimulation (TMS) | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT03698591/Prot_SAP_002.pdf
  • Informed Consent Form (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT03698591/ICF_003.pdf